CLINICAL TRIAL: NCT02568969
Title: Continuous Monitoring of Lactate in High-risk Cardiac Surgery
Brief Title: Lactate in High-risk Cardiac Surgery
Acronym: CLM-CARD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Northern State Medical University (Other)
Responsible Party: Principal Investigator, Mikhail Y. Kirov, Professor, Head of Anesthesiology Dept., Northern State Medical University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: LAC-1
Record Dates: First submitted 2015-09-30; First posted 2015-10-06 (Estimated); Last update posted 2016-03-24 (Estimated); Status verified 2016-03

CONDITIONS: Continuous Lactate Measurements; Cardiosurgery
Keywords: Cardiosurgery, lactate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Lactate monitoring (Experimental): The patients in the group will be subjected to the continuous perioperative monitoring of the venous blood lactate
  Interventions: Device: Eirus continuous lactate monitor

INTERVENTIONS:
Device: Eirus continuous lactate monitor — a triple-lumen central venous catheter (Eirus TLC) functioning as a regular central venous catheter (CVC) with an integrated microdialysis function will be inserted via the left jugular vein for continuous monitoring of lactate and glucose using Eirus intravascular microdialysis system (Maquet Critical Care, Solna, Sweden) after calibration with arterial sample. Eirus TLC will be used for both drug administration and blood sampling and will be removed postoperatively when a central line will no longer be necessary.
  Other Names: Eirus (Maquet)

SUMMARY:
The major combined interventions are between challenging and high-risk aspects of current cardiosurgical practice. The results of operation may be hampered by unexpected anatomic and technical features influencing the surgical approach as well as cardiopulmonary bypass (CPB), anesthesia, and respiratory support.

Plasma lactate concentration is a routine clinical indicator of the tissue oxygen shortage, and is routinely monitored in virtually all in-risk surgical and ICU patients. However, the discrete measurement of these values among with other biochemical values has a major drawback and continuous measurement can be beneficial.

The aim of our study is to assess the clinical usefulness and rationale for routine use of continuous monitoring of lactate in high-risk combined/complex cardiac surgery.

DETAILED DESCRIPTION:
The combination of coronary artery bypass grafting (CABG), repair of valve pathology and/or valve replacement remains a challenging and high-risk aspect of current cardiosurgical practice. Direct and indirect results of surgery are affected by the variety of factors including patient's age, general condition, preoperative severity of heart dysfunction and remodeling, etc. In addition, the results of operation may be hampered by unexpected anatomic and technical features influencing the surgical approach as well as duration of cardiopulmonary bypass (CPB) and aortic cross clamping, anesthesia, intensive care and respiratory support.

The combined and complex cardiac surgery requires CPB, which, in parallel with increased duration of intervention, induces systemic inflammatory response and ischemia-reperfusion injury. These pathophysiological mechanisms include activation of cytokines, complement, neutrophils, monocytes, endothelium and platelets. Neutrophil sequestration in the vital organs in response to chemotaxis and release of reactive oxygen species and inflammatory mediators may result in tissue hypoperfusion and multiple organ dysfunction syndrome, contributing to development of postoperative complications and adverse outcomes.

To alleviate CPB-induced systemic inflammatory response and organ-specific injury, different interventions exist, including meticulous hemodynamic and metabolic monitoring followed by goal-directed therapy. Several recent studies from our group and other authors have clearly demonstrated the beneficial effects of such an approach in cardiac surgery. In these settings, when the extraction of O2 on cellular level may be severely disturbed, the complex analysis of changes in tissue perfusion and oxygenation before adjusting the therapy may be useful.

Current technique of continuous monitoring of lactate using Eirus system has a potential to broaden our knowledge in this clinical scenario and reinforce a decision-making in high-risk cardiac surgery. Hence, continuous measurement of lactate may be a valuable adjunct to routine hemodynamic parameters and blood gases, facilitating changes in fluid therapy and inotrope/vasopressor support for the achievement an adequate balance between oxygen demand and delivery. Combination of continuously measured lactate with monitoring of cardiac output, mixed and central venous saturation and Pv-aCO2 seems to be an attractive approach to "global view" on the systemic oxygen transport at the bedside. Recently, the continuous monitoring of lactate has been validated in a pilot clinical study in cardiosurgical patients mostly with isolated CABG and aortic valve replacement with relatively short-term CPB, however its' role in combined cardiac surgery with prolonged CPB, representing the important setting for lactate-guided therapy, remains unsettled.

Thus, the aim of our study is to assess the use of continuous monitoring of lactate in high-risk combined/complex cardiac surgery.

ELIGIBILITY:
Inclusion Criteria:

* Informed consent.
* Age above 18 years.
* Presence of coronary artery disease and/or valve regurgitation and/or stenosis
* Elective complex (two and more valves) and combined (valve + CABG) cardiac surgery requiring CPB with expected duration > 90 min.

Exclusion Criteria:

* Participation in any other study.
* Morbid obesity (BWI > 40).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2015-03; Primary Completion 2015-11 (Actual); Study Completion 2015-11 (Actual)

PRIMARY OUTCOMES:
Hyperlactatemia | 0-24 hrs
  Presence of hyperlactatemia (> 2.0 mmol/l) in the intra- and postoperative period.

SECONDARY OUTCOMES:
Cardiac index | 0-24 hrs
  The incidence of low cardiac index (< 2,5 l/min/m2) The organ failure is to be diagnosed according to the well defined criteria
Acute kidney injury | 0-24 hrs
  The incidence of acute kidney injury according to KDIGO criteria
Respiratory distress | 0-24 hrs
  The incidence of acute respiratory distress syndrome (PaO2 / FiO2 < 300 mm Hg)

CONTACTS AND LOCATIONS:
Overall Officials: Mikhail Y. Kirov, MD, PhD, Principal Investigator — Northern State Medical State University
Locations (1):
- City hospital # 1 / Northern State Medical University,, Arkhangelsk, Russia